CLINICAL TRIAL: NCT03021772
Title: Efficacy of Neostigmine Versus Dexamethasone as Adjuvants to Lidocaine During Intravenous Local Anesthesia for Forearm Orthopedic Surgeries
Brief Title: Neostigmine Versus Dexamethasone as Adjuvants to Lidocaine During Intravenous Local Anesthesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MOHAMED F. MOSTAFA, Lecturer of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Bier Block
Record Dates: First submitted 2017-01-10; First posted 2017-01-16 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Adjuvants, Anesthesia
Keywords: Neostigmine; Dexamethasone; Intravenous Local Anesthesia
MeSH Terms: interventions — Neostigmine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group N (Active Comparator): 30 patients will receive intravenous 3mg/kg lidocaine 2 % (diluted with normal saline to 40 ml) + 0.5 mg neostigmine for Bier block.
  Interventions: Drug: Neostigmine
- Group D (Active Comparator): 30 patients will receive intravenous 3mg/kg lidocaine 2 % (diluted with normal saline to 40 ml) + 8 mg dexamethasone for Bier block.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Neostigmine — Patients will receive intravenous 3mg/kg lidocaine 2 % (diluted with normal saline to 40 ml) + 0.5 mg neostigmine for Bier block.
  Arms: Group N
Drug: Dexamethasone — Patients will receive intravenous 3mg/kg lidocaine 2 % (diluted with normal saline to 40 ml) + 8 mg dexamethasone for Bier block.
  Arms: Group D

SUMMARY:
Intravenous regional anesthesia (IVRA) is described firstly in 1908 by August Bier. It is simple, safe, reliable, less cost, efficient method in forearm surgery. The advantage of this method has fast return of motor and sensory function which enables patients for earlier discharge. However, this method has disadvantages such as tourniquet pain, insufficient muscle relaxation and postoperative analgesia.

Lidocaine inhibits action potential propagation within neuronal tissue by binding to receptors in Na+ channels located on the nerve cell membrane. Lidocaine IVRA is safe and effective and is associated with a rapid onset (4.5 minutes) of anesthesia after injection and termination of analgesia (5.8 ± 0.5 minutes) once the tourniquet is deflated.

Neostigmine is a typical cholinesterase inhibitor. It increases the level of acetylcholine (Ach) and indirectly stimulates both nicotinic and muscarinic receptors. In anesthesia, neostigmine is a drug that has been used for reversal of residual neuromuscular block. Administration of neostigmine by intrathecal and epidural routes has been found to cause analgesia by inhibition of the breakdown of Ach in the spinal cord.

Dexamethasone is commonly used in anesthesia to prevent postoperative nausea and vomiting (PONV). Two recent meta-analyses have documented that dexamethasone also reduced postoperative pain and opioid requirement. Intravenous dexamethasone has also been shown to improve postoperative pain control in patients receiving spinal or epidural morphine.

Hong et al reported that intravenous dexamethasone in combination with a caudal block with ropivacaine prolonged the duration of postoperative analgesia without adverse effects in children undergoing orchidopexy. So the investigators expect that addition of dexamethasone or neostigmine will affect duration and postoperative analgesia in bier block.

DETAILED DESCRIPTION:
This study will be a prospective clinical randomized controlled double-blind study using a computer-generated randomization. Neither the doctor "investigator" nor the participant "patient" will be aware of the group allocation or the drug used. The study drugs will be prepared by one of the supervisor anesthesiologists (not included in the procedure, observation or data collection).

The study will be carried out in Assiut University Hospital after approval from our local ethical committee.

Patients

The patients will be classified in two groups:

According to sample size calculator. Group D: will include 30 patients and will receive intravenous 3mg/kg lidocaine 2 % (diluted with normal saline to 40 ml) + 8 mg dexamethasone for bier block.

Group N: will include 30 patients and will receive intravenous 3mg/kg lidocaine 2 % (diluted with normal saline to 40 ml) + 0.5 mg neostigmine for bier block.

Methods

Before the procedure, the patient should be:

* Starved for 6-8 hours.
* Monitored closely (standard monitoring applied: HR, NIBP, SaO2 and RR)
* Adequately informed about the procedure and have consented to it.

The equipments required for IVRA include:

- Pneumatic tourniquet (checked for leaks before the procedure) and a pressure gauge.

* Esmarch bandage or Rhys-Davis exsanguination.
* Local anesthetic solution and the adjuvants.
* Resuscitation equipments and drugs.

Technique:

IVRA of the arm: a 22 G cannula is placed intravenously as distal as possible in the arm to be anesthetized. Venous access is established in the opposite arm to allow administration of fluids or other drugs if necessary. The double tourniquet (two tourniquets each 6 cm wide) or a single one (14 cm wide) is applied on the operated arm with generous layers of padding, ensuring that no wrinkles are formed and the tourniquet edges do not touch the skin.

The arm is exsanguinated either by using the Esmarch bandage or a Rhys-Davis exsanguinator. If this is impossible, exsanguination can be achieved by elevating the arm for 2-3 minutes while compressing the axillary artery. The distal tourniquet is inflated to at least 100 mm Hg higher than the patient's systolic blood pressure (250 - 300 mmHg). The proximal tourniquet is inflated to the same pressure.

After ensuring inflation, the distal cuff is deflated. Before injecting local anesthetic, it must be confirmed that no radial pulse is palpable. The local anesthetic is then injected slowly. A standard volume for injection into the upper limb is 40 ml, which can be increased to 50 ml in a fit, large adult.

If the injection is too rapid, the venous pressure may exceed the tourniquet pressure and the local anesthetic solution may escape into the systemic circulation. Surgical anesthesia is usually achieved within 15 minutes. The distal tourniquet, which overlies part of the anesthetized arm, can then be inflated and the proximal one deflated to relieve tourniquet pain. The cuff should not be deflated until 20 minutes after local anesthetic injection because systemic toxic doses of local anesthetic may occur.

Cuff deflation should be performed in cycles with deflation/inflation times of less than 10 seconds until the patient no longer exhibits signs of systemic toxicity (e.g. tingling of the lips, tinnitus or drowsiness). Therefore, the patient should be monitored closely for 30 minutes following tourniquet release. So, the investigators expect that addition of dexamethasone or neostigmine will affect duration and postoperative analgesia.

Data collection:

1. Patient's data: include patient's gender, age, weight, height, BMI and ASA classification.
2. Preoperative data:

   1. Basic Monitoring: heart rate (HR), non-invasive blood pressure (NIBP), arterial oxygen saturation (SaO2), respiratory rate (RR) will be recorded.
   2. Preoperative investigations: prothrombin time, prothrombin concentration and INR to avoid any risk of internal bleeding.
   3. Basal assessment of motor power and sensation of the limb:

<!-- -->

1. Motor power: Motor block was evaluated by thumb abduction (radial nerve), thumb adduction (ulnar nerve), thumb opposition (median nerve), and flexion at the elbow (musculocutaneous nerve) on a 3-point scale for motor function (0: normal motor function, 1: reduced motor strength but able to move fingers, 2: complete motor block).
2. Sensation: Sensory block (4 nerves) was assessed by ice packs using a 3-point scale: 0: normal sensation, 1: loss of sensation of cold (analgesia), 2: loss of sensation of touch (anesthesia).

   d- The standard value of visual analogue scale will be set as the score during passive exercise before the surgery.
3. Introperative data:

   1. Basic Monitoring: heart rate (HR), non-invasive blood pressure (NIBP), arterial oxygen saturation (SaO2), respiratory rate (RR) will be recorded every 10 minutes till the end of surgery.
   2. Sensory and motor block: Sensory and motor blocks will be evaluated every 5 minutes until 20 minutes after injection.

   Onset time will be defined as the time interval between the end of total local anesthetic administration and complete sensory block. Complete sensory block will be defined by anesthetic block (score 2) on all nerve territories.

   Complete motor block will be defined as absence of voluntary movement on hand and forearm (score 0).

   c- Duration of surgery.
4. Postoperative data:

   1. Duration of sensory and motor block:

      Duration of sensory block will be defined as the time interval between the end of local anesthetic administration and the complete resolution of anesthesia on all nerves.

      Duration of motor block will be defined as the time interval between the end of local anesthetic administration and the recovery of complete motor function of the hand and forearm.
   2. Duration of analgesia: interval between onsets of the block to the time of the first analgesic requirement.
   3. Analgesia assessment:

   Postoperatively, a Post-Anesthesia Care Unit (PACU) nurse will assess the quality of analgesia. The pain score will be recorded using the Visual Analouge Scale (VAS) 2, 4, 6, 12 and 24 hours after surgery. Significant pain is defined as one that has a score of ≥ 4 and as a consequence required a supplementary dose of analgesia. Intravenous Paracetamol 15 mg/kg, will be administered and recorded.

   d- Documentation of any complications: Includes local anesthetic toxicity & drug additives complications.

   Local anesthetic toxicity:

   • Initial symptoms are subjective and include perioral tingling or numbness, lightheadedness, tinnitus, metallic taste, slurred speech, auditory and visual disturbances.

   • Minor symptoms usually do not require treatment. If any of these occur observe patient closely and identify any potential reasons for systemic toxicity eg: check for cuff failure - re-inflate.
   * Significant neurotoxicity: Objective signs are usually excitatory: twitching, fasciculation and seizures:

     - Check for cuff failure - re-inflate immediately

     - Administer Midazolam 2.5-5.0 mg iv
     * Support the ABC's as indicated Most seizures are self-limiting but can be potentiated by hypoxia, acidosis and hypercarbia so these should be treated aggressively.
   * Significant cardiotoxicity: if occurs (eg: hypotension, bradycardia and arrhythmias):

   Give oxygen and adopt an ACLS approach Check for cuff failure - re-inflate immediately Bicarbonate may be indicated to address acidaemia.

   Drug additives complications:

   All patients will be monitored for any complications that may occur from any adjuvant drugs used in the study and will be treated promptly.

   Statistical analysis All data will be collected and analyzed using SPSS version 20 (SPSS, Inc., Chicago, Illinios, USA). Normally distributed data will be expressed as mean ± standard deviation, range, numbers and percentages. A probability (p) value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 - 60 years.
* ASA grade I - II.
* Surgical time does not exceed 90 minutes.

Exclusion Criteria:

* Patient refusal.
* Any contraindication of regional anesthesia block (e.g. Coagulopathy, infection at the needle insertion site or vascular insufficiency).
* A personal history of seizures, peripheral neurologic diseases, cardiac arrhythmias, sickle cell anemia, liver dis¬ease, renal dysfunction and cardiac conduction abnormalities.
* Patients with allergy to amide local anesthetics or medication included in the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Pain assessed on VAS | 24 hours
  perfalgan will be given when visual analogue score ≥ 4

SECONDARY OUTCOMES:
Sensory level | 2 hours
  duration of sensory block
Motor level | 2 hours
  duration of motor block
Number of patients with any complications | 24 hours
  Percentage of patients with any complications will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: HAMDY A. YOUSSEF, MD, Study Chair — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided